## **COVER PAGE**

## STATISTICAL ANALYSIS PLAN

OFFICIAL TITLE: Prognostic Relevance of Fatty Liver Disease for Patients With Chronic

Hepatitis B

**DATE OF DOCUMENT: December 31, 2021** 

## **Statistical Analysis Plan**

Data will be summarized using descriptive statistics. Quantitative variables will be compared between groups using standard parametric or non-parametric tests, and qualitative variables will be compared using the Chi-squared test. The cumulative probabilities of mortality or liver transplantation and liver-related complications will be estimated by the Kaplan-Meier method and compared by the log-rank test. Hazard ratios (HR) and 95% confidence interval (CI) estimates for the outcomes will be calculated by Cox proportional hazard model. All potential confounders, including age, sex, overweight/obese, diabetes, hypertriglyceridemia, hypertension, and statin use, will be considered for multivariable models to identify independent determinants of the study outcomes. Time at risk will be defined as the date of liver biopsy to the date of outcome or last follow-up. Statistical analyses will be done using SPSS version 18.0.